CLINICAL TRIAL: NCT04219202
Title: Neoadjuvant Irradiation of Retroperitoneal Soft Tissue Sarcoma With Ions Retro-Ion Prospektive Randomisierte Phase-II-Studie
Brief Title: Neoadjuvant Irradiation of Retroperitoneal Soft Tissue Sarcoma With Ions Retro-Ion
Acronym: Retro-Ion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Princip Investigator, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rad-ONK Retro-Ion
Record Dates: First submitted 2020-01-03; First posted 2020-01-06 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Sarcoma,Soft Tissue
MeSH Terms: conditions — Sarcoma | interventions — Proton Therapy; Heavy Ion Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proton Treatment (Active Comparator): Patient receive 39 Gy (in 13 fractions (SD 3,0 Gy) Proton Treatment
  Interventions: Radiation: Proton radiation
- Carbon Ion Treatment (Experimental): Patient receive 39 Gy (in 13 fractions (SD 3,0 Gy) Carbon Ion Treatment
  Interventions: Radiation: Carbon Ion radiation

INTERVENTIONS:
Radiation: Proton radiation — Therapeutic radiation Treatment with Protons
  Arms: Proton Treatment
Radiation: Carbon Ion radiation — Therapeutic radiation Treatment with Carbon Ions
  Arms: Carbon Ion Treatment

SUMMARY:
The study is a randomized, open, prospective phase II study. The aim of the study is to evaluate the safety and feasibility of a hypofractionated, accelerated radiation approach based on the incidence of grade 3-5 NCI Common Terminology Criteria for Adverse Events (NCI-CTC-AE ) toxicity and / or termination of the planned therapy for any reason with neoadjuvant radiation with active beam guidance of the retroperitoneal Sarcomas using protons or carbon ions before a subsequent tumor resection.

DETAILED DESCRIPTION:
With retroperitoneal sarcomas, the patient benefits from neoadjuvant radiotherapy. Due to the special physical properties of particles (protons and C12 carbon ions), in particular the steep lateral dose drop, an improved protection of adjacent risk organs is e.g. Intestine, kidneys, liver etc. during the process of applying radiotherapy is possible.

The primary study objective is to demonstrate the safety and conduct of study treatment and the incidence of Grade 3-5 NCI-CTC-AE toxicity and / or termination of preferred therapy for any reason. Further target parameter is the proportion of applied therapies without the occurance of degree 3-5 NCI-CTC-AE(s).

The patients are randomized 1: 1 into the two arms (carbon ions vs. protons). Patients receive 39 Gy in (SD 3.0 Gy) in 6 fractions per week.

Secondary study objectives are local control (LC), local progression-free survival from the start of therapy (LPFS), disease-free survival (DFS), overall survival (OS) and quality of life (QoL) determined according to the EORTC-Quality of Life Questionaire (QLQ)- C30 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed retroperitoneal soft-tissue sarcoma which is resectable or marginally resectable
* Karnofsky index of ≥ 70%
* Age from 18 years
* Completed patient information and written consent
* ability to give consent

Exclusion Criteria:

* Stage IV (distant metastases)
* Lymphogenic metastasis
* Metal implants at the level of the sarcoma, which influence the treatment planning
* Previous radiation therapy in the treatment area
* Desmoid tumors, peritoneal sarcomatosis, GIST
* Simultaneous participation in another clinical study that could influence the results of the respective study
* Active medical implants for which there is no license for ion irradiation at the time of treatment (e.g. pacemaker, defibrillator)
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-05-09 (Actual); Primary Completion 2026-05-09 (Estimated); Study Completion 2027-05-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of grad 3-5 NCI-CTC-AE toxicities | within 12 month after radiation treatment
  Evidence of the safety and practicability of the study treatment assessed for the incidence of grade 3-5 NCI-CTC-AE toxicity and / or termination of the planned therapy for any reason

SECONDARY OUTCOMES:
local Tumor control | within 12 month after radiation treatment
  Number of patients without new arising Tumors at the treated Tumor site
local Progression free survival | within 12 month after radiation treatment
  Number of patients without local Progression at the treated tumor site
disease free survival | within 12 month after radiation treatment
  Number of Patients without relapse of treated disease
Overall survival | within 12 month after radiation treatment
  Assesment of alive patients
Quality of live | within 12 month after radiation treatment
  Assessed by EORTC QLQ-C30, Minimum value 0; Maximum value 6

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Heidelberg, Radiation Oncology, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seidensaal K, Kieser M, Hommertgen A, Jaekel C, Harrabi SB, Herfarth K, Mechtesheimer G, Lehner B, Schneider M, Nienhueser H, Frohling S, Egerer G, Debus J, Uhl M. Neoadjuvant irradiation of retroperitoneal soft tissue sarcoma with ions (Retro-Ion): study protocol for a randomized phase II pilot trial. Trials. 2021 Feb 12;22(1):134. doi: 10.1186/s13063-021-05069-z. PMID 33579340